CLINICAL TRIAL: NCT00565006
Title: A Study to Investigate the Influence of MK0859 on Blood Pressure (MK-0859-012)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0859-012; 2007_656
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Ambulatory Blood Pressure
MeSH Terms: interventions — anacetrapib

INTERVENTIONS:
Drug: MK0859

SUMMARY:
This study will investigate the influence of MK0859 on ambulatory blood pressure, and how safe and tolerable MK0859 is on the subjects This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* You are between the ages of 45-75
* You are a man or non-pregnant woman
* You agree to not eat or drink fruit or fruit juices (orange, apple or grapefruit) for 2 weeks before starting study medication

Exclusion Criteria:

* You have smoked or used other nicotine-containing products (chewing tobacco) within the last 6 months
* You have used St. John's Wort or any products that include it within the last 2 weeks
* You have used herbal, organic, dietary or nutritional remedies within the last 2 weeks
* You have a history of drug allergies (anaphylaxis, angioedema)
* You have taken an investigational drug in another clinical trial within the last 4 weeks
* You have a history of cardiovascular disease including hypertension (high blood pressure)
* You have a history of renal disease
* You have a history of gall bladder disease or have had abnormal liver function tests
* You have a history of drug or alcohol abuse
* You drink more than 6 cups of caffeinated beverages a day (coffee, tea or cola)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-07; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Krishna R, Anderson MS, Bergman AJ, Jin B, Fallon M, Cote J, Rosko K, Chavez-Eng C, Lutz R, Bloomfield DM, Gutierrez M, Doherty J, Bieberdorf F, Chodakewitz J, Gottesdiener KM, Wagner JA. Effect of the cholesteryl ester transfer protein inhibitor, anacetrapib, on lipoproteins in patients with dyslipidaemia and on 24-h ambulatory blood pressure in healthy individuals: two double-blind, randomised placebo-controlled phase I studies. Lancet. 2007 Dec 8;370(9603):1907-14. doi: 10.1016/S0140-6736(07)61813-3. PMID 18068514